CLINICAL TRIAL: NCT06181890
Title: The Effect of Motivational Interviews Applied to Infertile Women on Infertility Affect, Self-Efficacy and Coping With Stress
Brief Title: The Effect of Motivational Interviews
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Kahramanmaras Sutcu Imam University (Other)
Responsible Party: Principal Investigator, Eda Sever, student, Kahramanmaras Sutcu Imam University
Other Study IDs: KSIU-SBF-ES-01
Record Dates: First submitted 2023-12-13; First posted 2023-12-26 (Actual); Last update posted 2023-12-26 (Actual); Status verified 2023-12

CONDITIONS: Infertility, Female
Keywords: Infertility; Motivational Interview; Stress
MeSH Terms: conditions — Infertility, Female; Infertility | interventions — Motivational Interviewing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- control group: Infertile women who will be included in the control group will be interviewed twice in total. Pretest data will be obtained by applying the "Personal Information Form", "Infertility Impact Scale", "Infertility Self-Efficacy Scale - Short Form" and "Coping with Infertility Stress Scale" in the first interview. Four weeks after obtaining the pre-test data, post-test data will be obtained by applying the "Infertility Impact Scale", "Infertility Self-Efficacy Scale - Short Form" and "Coping with Infertility Stress Scale".
- intervention group: Before starting motivational interviews with infertile women in the intervention group, pre-test data will be obtained by applying the "Personal Information Form", "Infertility Impact Scale", "Infertility Self-Efficacy Scale - Short Form" and "Coping with Infertility Stress Scale". A total of 4 sessions of motivational interviews will be held for infertile women, 1 session per week for four weeks. At the end of four weeks, post-test data will be obtained by applying the "Infertility Impact Scale", "Infertility Self-Efficacy Scale - Short Form" and "Coping with Infertility Stress Scale".
  Interventions: Other: Motivational Interview

INTERVENTIONS:
Other: Motivational Interview — The data of the research will be collected between October 2023 and June 2024. Each meeting will last approximately 15-30 minutes.
  Groups: intervention group

SUMMARY:
The aim of the study was to determine the effect of motivational interviews applied to infertile women on their ability to cope with infertility, self-efficacy and stress.

DETAILED DESCRIPTION:
There is no study in the literature on the effectiveness of motivational interviewing on being affected by infertility, self-efficacy and coping with stress. It is important for healthcare personnel to be easy to apply and short-term, to be aware of the effectiveness of the motivational interviewing technique, and to use this technique in communicating with the patient and changing behavior. Based on these, it was deemed necessary to examine the effect of motivational interviews for infertile women.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18 and over and have no problems communicating Those who have not previously or currently been diagnosed with a psychiatric disease Infertile women who volunteer will be included in the sample of the research

Exclusion Criteria:

* Pregnancy during the study, Having previously or currently participated in a motivational interviewing program, Those who want to leave the research, Not completing motivational interviewing sessions, Infertile women with any deficiencies or errors in any of the forms from which the data are obtained will be excluded from the sample.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Study Population: The population of the research will be infertile women who come to Kahramanmaraş Necip Fazıl City Hospital Gynecology and Pediatrics Annex Building for infertility treatment.
Sampling Method: Probability Sample
Enrollment: 84 (Estimated)
Dates: Start 2023-10-25 (Actual); Primary Completion 2024-06-25 (Estimated); Study Completion 2024-06-25 (Estimated)

PRIMARY OUTCOMES:
motivational interview | 1 month
  A total of 4 sessions of motivational interviews will be held for infertile women, 1 session per week for four weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Esra Karataş Okyay, Principal Investigator — Kahramanmaras Sutcu Imam University; Eda Sever, Study Director — Kahramanmaras Sutcu Imam University
Locations (1):
- Eda Sever, Kahramanmaraş, Onikişubat, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No